CLINICAL TRIAL: NCT03547440
Title: Determinants of Type 1 Diabetes (T1DM) Clinical Onset and Progression in Paediatric Immigrant Population
Brief Title: T1DM Clinical Onset and Progression in Paediatric Population
Acronym: Bioda
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Collaborators: Azienda Ospedaliero Universitaria Maggiore della Carita (Other); A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Deborah Traversi, Associate Professor, University of Turin, Italy
Other Study IDs: G12114000080001; RF-2011-02350617 (Other Grant/Funding Number: Italian Health Minister)
Record Dates: First submitted 2017-03-16; First posted 2018-06-06 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; immigrant; microbiota; bioindicator; Methanobrevibacter smithii
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — stool samples (from all the participants) and blood samples (only from T1DM) patients
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- type 1 diabetes mellitus: Children with type 1 diabetes mellitus, usually not obese, with diabetic ketoacidosis. They could be with or without stationary metabolic profile. They are recruited at the onset of the T1DM into the Torino and Novara Pediatric Hospitals and then they are divided in relation to the ethnicity.
- Control healthy: Healthy children without relevant metabolic or systemic co-morbility. They are recruited from orthopedy department of the Torino and Novara Pediatric hospitals and then they are divided in relation to the ethnicity

SUMMARY:
Diabetes Mellitus Type I is the chronic metabolic disease of childhood with the highest incidence in developed countries. Over the past 10 years the incidence of diabetes has been increased especially in immigrants children. The objective of the investigator's project is to evaluate factors that influence the T1DM course in immigrant and Italian children through an analysis of the relationship between socio-cultural determinants, lifestyles and metabolic control. The study population will consist of 100 children with first diagnosis of T1DM divided into two cohorts (Italian and immigrant children). The project consists in a follow-up of 18 months from first visit and will include laboratory tests, two questionnaires and determination of a microbiological indicator of the microbiota and levels of 25-hydroxyvitamin D. The research hypothesis is that the two groups of study population show a different metabolic control of diabetes due to differences in access to care, compliance to therapy and type of nutrition.

DETAILED DESCRIPTION:
Over the past ten years a contribution to the increasing incidence of T1DM is derived from children of foreign origin. As many studies confirmed environmental factors are involved in the onset and development of T1DM: type of nutrition, infections, perinatal events, characteristics of the microbial flora, 25-hydroxyvitamin D levels and early exposure to certain foods. Recent research has disclosed a tight connection between gut microbes, host metabolism and utilization and storage of energy. For this reason the microbiota could be implicated also into the diabetes ongoing. Methanobrevibacter smithii is the dominant methanogen in both the distal colon of individuals in health and disease. Some studies reported that immigrant children have a less efficient metabolic control in comparison to age-matched Italian children, thus identifying the different ethnic background as a risk factor for quality of life: a younger age at T1DM diagnosis is frequently observed in immigrant children, which may have also an increased risk of nutritional problems related to dietary habits, social disadvantage and poverty.

The project will make a comparative assessment in the two populations (italian and immigrant children). The research hypothesis is that the two analysed groups show a different metabolic control of diabetes due to differences in access to care, in compliance to therapy and in type of nutrition.

Specific Aim:

1. Estimate any discrepancies in the course of T1DM among the two populations by assessing the modality of hospital admission (ordinary or emergency) and the structures involved.
2. Evaluate the quantity range of a microbiological indicator of intestinal microbial flora, (Methanobrevibacter smithii) determined by molecular techniques on stool samples and the levels of 25-hydroxyvitamin D in serum. That difference will be evaluated on immigrants and non-immigrants diabetic children and on a control group of healthy children.
3. Estimate of the main outcomes of two T1DM populations (glycated hemoglobin, number of hospitalizations for acute events with the calculation of hospital days per year, U insulin / kg / day, dose of C-peptide as an expression of residual pancreatic function) and their compliance to therapy and prescriptions (frequency of tests and visits, adherence to insulin therapy, dietary lifestyles).

Case-control at the onset of Italian T1DM versus Immigrant T1DM by assessing hospital admissions [Aim 1]

Origin-stratified case control [Case (T1DM) vs double control (healthy), italian and immigrant: evaluation microbiota/metabolic profile, vit D] [Aim 2]

Prospective cohort study (TDM1 italian vs TDM1 immigrant: evaluation of the impact of social and health-related factors) [Aim 3]

ELIGIBILITY:
Inclusion Criteria:

1. Cases migrants : T1DM's recent diagnosis
2. Italian cases : comparable to individual characteristics, living area, mainly age and gender
3. Controls: healthy children (two control comparable for each case)

Exclusion Criteria:

1. Children with parents of mixed origin
2. Children with chronic gastrointestinal disorders (such as irritable bowel syndrome) or other relevant metabolic or systemic co-morbility
3. Children who used antibiotics or with diarrhea in the last 15 days

Max Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children living in the Piedmont region. Primary care clinic of Torino and Novara (diabetologia for cases and orthopedia and general population for controls)
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2015-03-18 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-09-18 (Actual)

PRIMARY OUTCOMES:
Metabolic control | at onset
  The blood pH of the patients are measured at the onset to define ketoacidosis following normal standard hospital procedure.

SECONDARY OUTCOMES:
Body mass index | at onset
  calculated as (weight (kg))/(height (meters))exp2
Glycated hemoglobin | at onset
  in % and as mmol/mol
Diet behaviour | at onset
  The 24h-recall technique reconstructed meals and food intake on a recent "typical" day, estimating, under a bromatology point of vie, inputs according to food composition database for epidemiological studies in Italy (BDA)
vitamin D | at the onset
  evaluated from serum sample as 25-hydroxyvitamin D (ng/ml)
Microbiome bioindicators | at onset
  The Denaturing Gradient Gel Electrophoresis profile was evaluated for each patients starting from the stool sample. Shannon index is calculated (theory range from 0 to infinite; in literature from 0.1 to 4)
Methanobrevibacter smithii | at onset
  Starting from the stool DNA extracted, following bioindicator measured by quantitative Real Time Polymerase Chain Reaction: Methanobrevibacter smithii (num gene copies - both as 16S ribosomal RNA gene and nifH gene /g stool)
Akkermansia muciniphila quantification in stool | at onset
  Starting from the stool DNA extracted, following bioindicator measured by quantitative Real Time Polymerase Chain Reaction : Akkermansia muciniphila (num copies 16SrDNA /g stool)

OTHER OUTCOMES:
Metabolic control 2 | at onset
  The blood carbonate of the patients are measured at the onset to define ketoacidosis

CONTACTS AND LOCATIONS:
Overall Officials: Roberta T Siliquini, Prof., Principal Investigator — University of Turin - Hygiene and Preventive Medicine
Locations (3):
- Italy (3):
  - Pediatric Clinic - Hospital "Maggiore della Carità" of Novara, Novara
  - Dept. of Public Health and Pediatrics, Torino
  - Dep. of Medicine Science, Turin

IPD SHARING:
Plan to Share IPD: No